CLINICAL TRIAL: NCT02416804
Title: Postoperative Analgesia With Buprenorphine Transdermal System (BTDS) Versus Tramadol for Postoperative Pain Control and Quality of Life After Spinal Surgery
Brief Title: Postoperative Analgesia With Buprenorphine for Postoperative Pain Control and Quality of Life After Spinal Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin S. Yeom, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BTDS_001
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Spinal Stenosis; Pain, Postoperative
Keywords: buprenorphine; transdermal system; Pain, postoperative; Quality of life; Spinal stenosis; Posterior lumbar fusion
MeSH Terms: conditions — Spinal Stenosis; Pain, Postoperative | interventions — Buprenorphine; Tramadol

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Buprenorphine (Experimental): Buprenorphine group : They will apply 3 days after the spine operation.
  Interventions: Drug: Buprenorphine
- Tramadol (Active Comparator): Tramadol group : They will take a pill of tramadol analgesics.
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Buprenorphine — Buprenorphine transdermal patch Initial : 5 μg/hr Sequential increasing of dose : 5 μg/hr -> 10 μg/hr -> 15 (5+10) μg/hr -> 20 μg/hr
  Other Names: Norspan
  Arms: Buprenorphine
Drug: Tramadol — Tramadol Initial : 150 mg/d Sequential increasing of dose : 150 mg/d -> 200 mg/d -> 250 mg/d -> 300 mg/d
  Other Names: Zytram
  Arms: Tramadol

SUMMARY:
Major purpose of this research is to evaluate the effect and usefulness of Buprenorphine transdermal system (MTDS) among the patients with lumbar spinal disease who was performed the single-level posterior lumbar fusion.

After surgery, all the patients apply the patient-controlled analgesia. After three days of surgery, patients are divided into two groups.Group A is an experimental group that administer the BTDS after surgery, and Group B is a control group that take tramadol analgesics. If the patient's pain score exceeds the NRS 4, they can take the additional rescue medicine, acetaminophen.

After the surgery, patient's pain score and quality of life would be recorded sequentially. The time of recording is postoperative 36 hours, 72 hours, 7 days, 2 weeks, 4 weeks, and 3 months, respectively.

ELIGIBILITY:
Inclusion Criteria:

* adults over 20 years
* taking the lumbar spinal surgery : single-level, posterior fusion
* stay in hospital more than 2 days after operation

Exclusion Criteria:

* pregnancy or breast-feeding
* allergy or contraindication to buprenorphine
* patient with decreased lung function
* patient with taking MAO inhibitor or anticonvulsant
* patient with brain lesion, or severe liver disease
* dependence in opioid drugs
* taking muscle relaxant or tranquilizer
* patient had taken buprenorphine preoperatively
* taking strong opioids before enrolling the study
* another severe source of pain except lumbar spine
* severe cardiovascular, pulmonary, or renal compromised patients

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2015-01 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Pain intensity score : pain NRS scale | 3 months
  We will estimate pain NRS scale at 36 hours, 72 hours, 7 days, 2 weeks, 4 weeks, and 3 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Joong Kim, MD, Study Director — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim HJ, Ahn HS, Nam Y, Chang BS, Lee CK, Yeom JS. Comparative study of the efficacy of transdermal buprenorphine patches and prolonged-release tramadol tablets for postoperative pain control after spinal fusion surgery: a prospective, randomized controlled non-inferiority trial. Eur Spine J. 2017 Nov;26(11):2961-2968. doi: 10.1007/s00586-017-5213-5. Epub 2017 Jul 20. PMID 28730328